CLINICAL TRIAL: NCT04759820
Title: A Multicentre Randomized Controlled Clinical Study of the Efficacy of Carbon Nanoparticles Versus Indocyanine Green in Surgical Treatment of Colorectal Cancer
Brief Title: Carbon Nanoparticles vs Indocyanine Green
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LI XIN-XIANG (Other)
Responsible Party: Sponsor-Investigator, LI XIN-XIANG, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRC-SH02
Record Dates: First submitted 2021-02-07; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Number of Lymph Node Retrieved

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nano carbon group (Experimental): Injection of carbon nanoparticle
  Interventions: Drug: injecting Carbon Nanoparticles Suspension
- Indocyanine green group (Active Comparator): Injection of indocyanine green
  Interventions: Drug: Injecting indocyanine green

INTERVENTIONS:
Drug: injecting Carbon Nanoparticles Suspension — injecting Carbon Nanoparticles Suspension for lymph node detection
  Arms: Nano carbon group
Drug: Injecting indocyanine green — Injecting indocyanine green for lymph node detection
  Arms: Indocyanine green group

SUMMARY:
Both nano carbon and ICG as lymph node tracers in colorectal cancer have their own value, this study was to contrast two tracers in colorectal cancer surgeries, so as to find out the best lymphnode tracer in colorectal cancer, in order to further improve postoperative lymph node inspection, precise postoperative adjuvant therapy and improve the patients' long-term survival.

ELIGIBILITY:
Inclusion Criteria:

1. Colorectal cancer was confirmed by preoperative fibrocolonoscopy and pathological examination;
2. The operative requirements of the patients included in the study: laparoscopic radical surgery of colon/rectal cancer, indocyanine green group should be used fluorescent laparoscopic (Pinpoint) surgery;
3. The lower edge of the lesion is located more than 10cm from the anus;
4. Age 18 ~ 70;
5. The results of laboratory examination before enrollment met the following surgical conditions: neutrophils (ANC) ≥1.5×109/L, platelets (PLT) ≥ 100×109/L, total bilirubin (TBI) ≤1.5× upper limit of normal (2mg/ dL), alanine aminotransferase (ALT), ascarate aminotransferase (AST) ≤2× upper limit of normal;The coagulation parameters were in the normal range.
6. Patients had no psychological, family, social, or geographical constraints that affected protocol compliance and follow-up time
7. Patient signs informed consent;

Exclusion Criteria:

1. Under 18 years old or above 70 years old;
2. Other types of colorectal cancer (adenosquamous cell carcinoma, squamous cell carcinoma, neuroendocrine tumor, clear cell carcinoma, spindle cell carcinoma, undifferentiated carcinoma)
3. Rectum cancer less than 10cm from the anus;
4. Previous abdominal surgery;
5. Neoadjuvant therapy was received preoperatively, including radiotherapy and chemotherapy;
6. Due to various reasons, preoperative colonoscopic injection of carbon nanoparticles/indocyanine green labeling was not possible;
7. Intraoperative radical surgery cannot be performed due to various reasons;
8. Acute abdomen: intestinal obstruction, intestinal wringing, peritonitis, etc.;
9. Combined with other site metastasis;
10. Have severe heart, lung, liver and kidney diseases and cannot tolerate surgery;
11. Active stage of liver disease or abnormal liver function, ALT, AST, TBIL more than twice the upper limit of normal value;
12. Renal function impairment, Cr≥2 times the upper limit of normal or BUN≥2 times the upper limit of normal;
13. The subjects' white blood cells are lower than the lower limit of normal value, or their platelets are lower than the lower limit of normal value, or have other diseases of the blood system;
14. People with mental illness or mental retardation who cannot describe their feelings correctly;
15. Severe disorder of coagulation mechanism and bleeding tendency;
16. Have a history of serious uncontrolled medical disease or recent myocardial infarction (within 3 months);Acute infection;
17. Patients with uncontrolled severe hypertension and severe diabetes after intervention treatment;
18. Allergic to the test drug;
19. A history of alcohol, drug or substance abuse;
20. Participants who had participated in any drug trial within 3 months prior to enrollment;
21. Other subjects considered by the researcher to be unsuitable for inclusion in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of lymph nodes detected | 1 week after surgery
Number of positive lymph nodes detected at different T stages | 1 week after surgery
the ratio of positive lymph nodes | 1 week after surgery

SECONDARY OUTCOMES:
patients' Disease-Free Survival(DFS) | 1 year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China